CLINICAL TRIAL: NCT06450626
Title: Introduction of a Music-based Intervention for Patients Receiving Infusions at the Lifespan Cancer Institute Infusion Center in the Miriam Hospital
Brief Title: Music Therapy at TMH Infusion Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: The Warren Alpert Medical School of Brown University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00000448
Record Dates: First submitted 2024-05-31; First posted 2024-06-10 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Music Therapy
Keywords: Chemotherapy; Infusion Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Listening Music Intervention (Experimental): Participants listen to 30 minutes of a music playlist of their choice.
  Interventions: Other: Listening Music Intervention

INTERVENTIONS:
Other: Listening Music Intervention — Participants will listen to a music playlist while vitals are monitored, along with completing a pre- and post-assessment survey (both of which are the Edmonton Symptom Assessment Scale). Participants will also be asked a set of qualitative questions about their overall experience with the music therapy session.

SUMMARY:
The goal of this clinical trial is to test the effects of a listening music intervention on the symptom burden carried by patients who are receiving infusions at the Lifespan Cancer Institute of Miriam Hospital in Providence, Rhode Island. The main questions it aims to answer are:

* Will a music therapy intervention help reduce physical and mental symptom burden?
* Will a music therapy intervention be beneficial on physiological parameters during the infusion sessions, such as heart rate, respiratory rate, and blood rate?

Participants will undergo the following main tasks:

* Prior to the infusion, participants will be given a pre-assessment survey reflecting on their previous experiences with infusions.
* During the infusion, participants will listen to a self-selected playlist either on their own device or on an iPad provided by the clinic, and vitals will be monitored.
* After the session, participants will be given a post-assessment survey to evaluate outcomes of the intervention.
* Participants will also be asked a set of qualitative questions about their overall experience with the music therapy session.

DETAILED DESCRIPTION:
An estimated 17 million Americans are living with cancer, and the majority receive chemotherapy annually, which, in addition to common side effects like pain, fatigue, nausea, vomiting, and hair loss, also imposes a significant psychological and emotional toll on patients. Studies consistently show a high prevalence of depression and anxiety among cancer patients due to both the disease and the therapeutic burden, with prolonged chemotherapy being a particularly significant risk factor. This underscores the need for nonpharmacological and non-invasive treatments to reduce the negative emotional states, psychological burden, and stress that often accompany chemotherapy. Music therapy has increasingly been utilized in clinical settings as a complementary intervention, benefiting various populations, including those with dementia-related disorders, by treating cognitive and behavioral symptoms through social interaction and other acute benefits. Passive music therapy, such as listening to recorded or live music, has been shown to ease psychosocial symptoms, even in the absence of a trained music therapist. Overall, music therapy promotes wellness, manages stress, alleviates pain, enhances memory, improves communication, and supports physical rehabilitation. For instance, in hypertensive young adults, four weeks of passive music therapy significantly lowered systolic blood pressure and heart rate, suggesting a soothing and rehabilitative effect. Additionally, singing along to music boosts cytokine levels, indicating strengthened immunity through improved mood and reduced stress. Music therapy research supports its benefits for cancer patients, as studies have shown improved mood, reduced distress, increased resilience, and decreased anxiety and heart rate during chemotherapy. Despite these demonstrated benefits, music therapy services are under-resourced, particularly in Rhode Island, where only one licensed music therapist was reported in 2020, serving around 2000 clients across eight facilities. This project aims to implement a music therapy program at Miriam Hospital to enhance the well-being of chemotherapy patients and potentially expand to other Lifespan Infusion Centers in Rhode Island, such as Rhode Island Hospital and Newport Hospital. Given the lack of structured music therapy programs for oncology patients in Rhode Island, this initiative seeks to establish a formal music therapy offering at Miriam Hospital, setting the stage for broader adoption and integration of music therapy in cancer care across the state.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient hearing capacity to hear music
* Scheduled for a chemotherapy infusion lasting at least 30 minutes
* Ability to complete pre- and post-assessments in English

Exclusion Criteria:

* Participants who have had a prior infusion session with a music therapy intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-06-19 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Effect of Music Listening Intervention on Common Symptoms Among Patients with Advanced Cancer via the Edmonton Symptom Assessment Scale | Baseline and 30 minutes (after the music listening intervention)
  The Edmonton Symptom Assessment Scale (ESAS) is now commonly used for symptom screening and longitudinal monitoring in patients seen by palliative care, oncology, nephrology, and other disciplines in both inpatient and outpatient settings. The ESAS is also a valid and reliable tool to assist in the assessment of nine common symptoms experienced by cancer patients. Possibles scores for each symptom range from 0 (no symptom feeling) to 10 (worst symptom feeling)
Change from Baseline in Heart Rate After Music Listening Intervention | Baseline and 30 minutes (after the music listening intervention)
  Heart rate is a physiological vital sign that is routinely taken by nurses before and after infusion sessions but is also a useful indicator of overall health status and relaxation. Heart rate will be measured in heart beats per minute.
Change from Baseline in Respiratory Rate After Music Listening Intervention | Baseline and 30 minutes (after the music listening intervention)
  Respiratory rate is a physiological vital sign that is routinely taken by nurses before and after infusion sessions but is also a useful indicator of overall health status and relaxation. Respiratory rate will be measured in breaths at rest per minute.
Change from Baseline in Blood Pressure After Music Listening Intervention | Baseline and 30 minutes (after the music listening intervention)
  Blood pressure is a physiological vital sign that is routinely taken by nurses before and after infusion sessions but is also a useful indicator of overall health status and relaxation. Blood pressure will be measured in mmHg.
Qualitative Satisfaction Level After Music Listening Intervention | Baseline and 30 minutes (after the music listening intervention)
  Vetted questions with the study director, Dr. Fred Schiffman, serve to measure participant satisfaction with the music listening intervention and if the experience improved their hospital stay. The questions also ask participants to reflect on any pieces of music that particularly connected with them during their infusion experience and why.
  These questions are qualitative in nature so there are no associated scales nor minimum and maximum values.

CONTACTS AND LOCATIONS:
Overall Officials: Fred J Schiffman, MD, Study Director — Brown University; Diana A Wang, BA, Principal Investigator — Brown University; Claire Lin, BA, Principal Investigator — Brown University; Ishaani Khatri, BA, Principal Investigator — Brown University
Locations (1):
- Lifespan Cancer Institute at The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers. All collected data will be kept internal to researchers on the project.

REFERENCES:
- [Derived] Khatri IS, Wang D, Lin C, Schiffman F, Guyer D. Infusion of Sound: Personalized Receptive Music-Based Intervention (rMBI) During Infusion Sessions. J Palliat Med. 2025 Dec 12. doi: 10.1177/10966218251406793. Online ahead of print. PMID 41467890

DOCUMENTS (1):
  • Study Protocol (2024-05-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT06450626/Prot_000.pdf